CLINICAL TRIAL: NCT02421510
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of LX4211 as Adjunct Therapy in Adult Patients With Type 1 Diabetes Mellitus Who Have Inadequate Glycemic Control With Insulin Therapy
Brief Title: Efficacy, Safety, and Tolerability Study of Sotagliflozin as Adjunct Therapy in Adult Patients With Type 1 Diabetes Mellitus Who Have Inadequate Glycemic Control With Insulin Therapy
Acronym: inTandem2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-310-T1DM; LX4211.310 (Other: Lexicon Pharmaceuticals); 2014-005153-39 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: High level of sugar (glucose) in the blood
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Two placebo-matching sotagliflozin tablets, once daily, orally, before the first meal of the day for 24 weeks followed by a 28-week extension period.
  Interventions: Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Sotagliflozin 200 milligram (mg) (one 200 mg tablet and one placebo tablet), once daily, orally, before the first meal of the day for 24 weeks followed by a 28-week extension period.
  Interventions: Drug: Sotagliflozin
- Sotagliflozin 400 mg (Experimental): Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, before the first meal of the day for 24 weeks followed by a 28-week extension period.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — High dose Sotagliflozin, once daily, before the first meal of the day
  Arms: Sotagliflozin 400 mg
Drug: Sotagliflozin — Low dose Sotagliflozin,once daily, before the first meal of the day
  Arms: Sotagliflozin 200 mg
Drug: Placebo — Placebo, once daily, before the first meal of the day
  Arms: Placebo

SUMMARY:
This Phase 3 study was intended to demonstrate superiority of either Sotagliflozin high dose or low dose versus placebo on glycosylated hemoglobin A1C (A1C) reduction at Week 24 when used as an adjunct in adult participants with type 1 diabetes mellitus (T1D) who have inadequate glycemic control with insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant who gave written informed consent to participate in the study in accordance with local regulations.
* Adult participants 18 years and older with a diagnosis of T1D made at least 1 year prior to informed consent.
* Participants treated with insulin or insulin analog delivered via continuous subcutaneous insulin infusion (CSII) or multiple daily injections (MDI).
* Willing and were able to perform Self-monitoring of blood glucose (SMBG) and completed the study diary as required per protocol.
* At the Screening Visit, A1C was between 7.0% to 11.0%.
* Females of childbearing potential must use an adequate method of contraception and have a negative pregnancy test.

Exclusion Criteria:

* Use of antidiabetic agent other than insulin or insulin analog at the time of screening.
* Use of sodium-glucose cotransporter (SGLT) inhibitors within 8 weeks prior to screening.
* Chronic systemic corticosteroid use.
* Type 2 diabetes mellitus (T2DM), or severely uncontrolled T1D as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sawhney, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (78):
- Austria (2):
  - Lexicon Investigational Site, Linz
  - Lexicon Investigational Site, Vienna
- Belgium (5):
  - Lexicon Investigational Site, Antwerp
  - Lexicon Investigational Site, Brussels
  - Lexicon Investigational Site, Edegem
  - Lexicon Investigational Site, Leuven
  - Lexicon Investigational Site, Sint-Niklaas
- Bulgaria (6):
  - Lexicon Investigational Site, Lovech
  - Lexicon Investigational Site, Plovdiv
  - Lexicon Investigational Site, Rousse
  - Lexicon Investigational Site, Smolyan
  - Lexicon Investigational Site, Sofia
  - Lexicon Investigational Site, Varna
- France (4):
  - Lexicon Investigational Site, Béziers
  - Lexicon Investigational Site, Dijon
  - Lexicon Investigational Site, Nantes
  - Lexicon Investigational Site, Nîmes
- Germany (6):
  - Lexicon Investigational Site, Düsseldorf
  - Lexicon Investigational Site, Hamburg
  - Lexicon Investigational Site, Hanover
  - Lexicon Investigational Site, Mainz
  - Lexicon Investigational Site, Münster
  - Lexicon Investigational Site, Neuwied
- Hungary (4):
  - Lexicon Investigational Site, Budapest
  - Lexicon Investigational Site, Gyula
  - Lexicon Investigational Site, Hódmezővásárhely
  - Lexicon Investigational Site, Zalaegerszeg
- Israel (7):
  - Lexicon Investigational Site, Haifa
  - Lexicon Investigational Site, Holon
  - Lexicon Investigational Site, Jerusalem
  - Lexicon Investigational Site, Petah Tikva
  - Lexicon Investigational Site, Tel Aviv
  - Lexicon Investigational Site, Tel Litwinsky
  - Lexicon Investigational Site, Ẕerifin
- Italy (6):
  - Lexicon Investigational Site, Catania
  - Lexicon Investigational Site, Milan
  - Lexicon Investigational Site, Palermo
  - Lexicon Investigational Site, Perugia
  - Lexicon Investigational Site, Pisa
  - Lexicon Investigational Site, Roma
- Lithuania (2):
  - Lexicon Investigational Site, Jonava
  - Lexicon Investigational Site, Kaunas
- Lexicon Investigational Site, Dordrecht, Netherlands
- Poland (7):
  - Lexicon Investigational Site, Katowice
  - Lexicon Investigational Site, Krakow
  - Lexicon Investigational Site, Lodz
  - Lexicon Investigational Site, Lublin
  - Lexicon Investigational Site, Poznan
  - Lexicon Investigational Site, Szczecin
  - Lexicon Investigational Site, Warsaw
- Romania (7):
  - Lexicon Investigational Site, Bacau
  - Lexicon Investigational Site, Bucharest
  - Lexicon Investigational Site, Buzău
  - Lexicon Investigational Site, Galati
  - Lexicon Investigational Site, Oradea
  - Lexicon Investigational Site, Sibiu
  - Lexicon Investigational Site, Târgu Mureş
- Slovakia (5):
  - Lexicon Investigational Site, Bratislava
  - Lexicon Investigational Site, Košice
  - Lexicon Investigational Site, Nové Zámky
  - Lexicon Investigational Site, Štúrovo
  - Lexicon Investigational Site, Vrútky
- Spain (5):
  - Lexicon Investigational Site, Barcelona
  - Lexicon Investigational Site, Granada
  - Lexicon Investigational Site, Málaga
  - Lexicon Investigational Site, Seville
  - Lexicon Investigational Site, Valencia
- Sweden (3):
  - Lexicon Investigational Site, Härnösand
  - Lexicon Investigational Site, Kristianstad
  - Lexicon Investigational Site, Stockholm
- Lexicon Investigational Site, Sankt Gallen, Switzerland
- United Kingdom (7):
  - Lexicon Investigational Site, Birmingham
  - Lexicon Investigational Site, Blackburn
  - Lexicon Investigational Site, Bristol
  - Lexicon Investigational Site, Glasgow
  - Lexicon Investigational Site, Leeds
  - Lexicon Investigational Site, Leicester
  - Lexicon Investigational Site, Sheffield

REFERENCES:
- [Derived] Peters AL, McGuire DK, Danne T, Kushner JA, Rodbard HW, Dhatariya K, Sawhney S, Banks P, Jiang W, Davies MJ, Lapuerta P. Diabetic Ketoacidosis and Related Events With Sotagliflozin Added to Insulin in Adults With Type 1 Diabetes: A Pooled Analysis of the inTandem 1 and 2 Studies. Diabetes Care. 2020 Nov;43(11):2713-2720. doi: 10.2337/dc20-0924. Epub 2020 Sep 14. PMID 32928957
- [Derived] Danne T, Joish VN, Afonso M, Banks P, Sawhney S, Lapuerta P, Davies MJ, Buse JB, Lin D, Reaney M, Guillonneau S, Snoek FJ, Bailey TS, Polonsky WH. Improvement in Patient-Reported Outcomes in Adults with Type 1 Diabetes Treated with Sotagliflozin plus Insulin Versus Insulin Alone. Diabetes Technol Ther. 2021 Jan;23(1):70-77. doi: 10.1089/dia.2020.0068. PMID 32721228
- [Derived] Ervin C, Joish VN, Evans E, DiBenedetti D, Reaney M, Preblick R, Castro R, Danne T, Buse JB, Lapuerta P. Insights Into Patients' Experience With Type 1 Diabetes: Exit Interviews From Phase III Studies of Sotagliflozin. Clin Ther. 2019 Nov;41(11):2219-2230.e6. doi: 10.1016/j.clinthera.2019.09.003. Epub 2019 Oct 3. PMID 31587812
- [Derived] Danne T, Cariou B, Buse JB, Garg SK, Rosenstock J, Banks P, Kushner JA, McGuire DK, Peters AL, Sawhney S, Strumph P. Improved Time in Range and Glycemic Variability With Sotagliflozin in Combination With Insulin in Adults With Type 1 Diabetes: A Pooled Analysis of 24-Week Continuous Glucose Monitoring Data From the inTandem Program. Diabetes Care. 2019 May;42(5):919-930. doi: 10.2337/dc18-2149. Epub 2019 Mar 4. PMID 30833371
- [Derived] Danne T, Cariou B, Banks P, Brandle M, Brath H, Franek E, Kushner JA, Lapuerta P, McGuire DK, Peters AL, Sawhney S, Strumph P. HbA1c and Hypoglycemia Reductions at 24 and 52 Weeks With Sotagliflozin in Combination With Insulin in Adults With Type 1 Diabetes: The European inTandem2 Study. Diabetes Care. 2018 Sep;41(9):1981-1990. doi: 10.2337/dc18-0342. Epub 2018 Jun 24. PMID 29937431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 96 investigative sites throughout 17 countries from 21 May 2015 to 23 June 2017.
Pre-assignment Details: 995 participants were screened and 782 participants with a diagnosis of Type 1 diabetes mellitus were randomized equally in 1 of 3 treatment groups: sotagliflozin 400 mg, sotagliflozin 200 mg or placebo.
Groups:
- Sotagliflozin 200 mg: Sotagliflozin 200 mg (one 200 mg tablet and one placebo tablet), once daily, orally, before the first meal of the day for 24 weeks followed by a 28-week extension period.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 258 | 261 | 263
Completed the 24 Week Treatment Period | 236 | 239 | 240
Completed (Participants who completed 52 week treatment (24 weeks + 28 extension weeks) period.) | 225 | 226 | 227
Not Completed | 33 | 35 | 36
Not completed — Other | 4 | 2 | 3
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Noncompliance with study drug | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 3
Not completed — Adverse Event | 9 | 10 | 18
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 18 | 12
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis included participants from the modified intent to treat (mITT) population, which included all randomly assigned participants who had taken at least 1 dose of study drug, analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 258 | 261 | 263 | 782
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (13.42) | 42.3 (13.59) | 41.7 (13.23) | 41.2 (13.44)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 244 | 252 | 253 | 749
  From 65-84 years | 14 | 9 | 10 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 122 | 130 | 376
  Male | 134 | 139 | 133 | 406
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 250 | 252 | 250 | 752
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 10 | 23
Insulin Delivery Method [Count of Participants; unit: Participants]
  Continuous Subcutaneous Insulin Infusion (CSII) | 66 | 68 | 67 | 201
  Multiple Daily Injections (MDI) | 192 | 193 | 196 | 581
Hemoglobin A1C (A1C) [Count of Participants; unit: Participants]
  <= 8.5% | 200 | 203 | 204 | 607
  >8.5% | 58 | 58 | 59 | 175
Hemoglobin A1C Value at Actual Week -2 Value [Count of Participants; unit: Participants] — Some sites entered the wrong Week -2 A1C stratum for some participants at randomization. This value is based on the stratum, participants should have been categorized based on their actual Week -2 A1C value.
  Participants
    <= 8.5% | 202 | 205 | 208 | 615
    >8.5% | 56 | 56 | 55 | 167
Body Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 81.08 (16.857) | 81.93 (17.386) | 81.97 (17.963) | 81.66 (17.394)
Duration of Diabetes [Mean (Standard Deviation); unit: Years] | 18.1 (10.72) | 18.2 (10.82) | 18.9 (11.18) | 18.4 (10.90)
Daily Total Insulin Dose [Mean (Standard Deviation); unit: International units per kilogram (IU/kg)] | 0.75 (0.295) | 0.73 (0.277) | 0.74 (0.267) | 0.74 (0.280)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. Least square (LS) means were obtained from a mixed-effects model for repeated measures (MMRM) that included fixed, categorical effects of treatment, randomization strata of insulin delivery method (MDI, CSII), randomization strata of Week -2 A1C (<= 8.5%, >8.5%), time (study week), a treatment-by-time interaction, and baseline A1C-by-time interaction as a covariate. A negative change from baseline (a reduction of A1C value at Week 24) indicates an improvement.
Time Frame: Baseline to Week 24
Population: Analysis included participants from the modified intent to treat (mITT) population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of A1C
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 239 | 239 | 241
Percentage of A1C | -0.02 (0.044) | -0.39 (0.044) | -0.37 (0.043)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline A1C-by-time interaction as a covariate; Test type: Superiority; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -0.37, 95% CI 2-sided [-0.48 to -0.25], Standard Error of Mean 0.058 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; LS means and p-values were obtained from Mixed effect Model Repeat Measurement (MMRM) model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline A1C- by-time interaction as a covariate; Test type: Superiority; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -0.35, 95% CI 2-sided [-0.47 to -0.24] — Sotagliflozin 400 mg versus Placebo

2. Secondary Outcome: Percentage of Participants With A1C <7.0% at Week 24 and no Episode of Severe Hypoglycemia, and no Episode of Diabetic Ketoacidosis (DKA) From Baseline to Week 24
Description: The composite endpoint included blood samples for the assessment of Hemoglobin A1C to determine the participants with a value <7.0% and a central blinded adjudication process to determine whether participants experienced either DKA or severe hypoglycemia. Only positively adjudicated severe hypoglycemia and diabetic ketoacidosis were included in the analysis.
Time Frame: Baseline to Week 24
Population: Analysis included participants from the mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 258 | 261 | 263
Percentage of participants | 15.1 | 31.4 | 32.3
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; P-values were obtained from a Cochran-Mantel-Haenszel (CMH) test stratified by the different levels of the randomization stratification factors of insulin delivery method (MDI, CSII) and Week -2 A1C (<=8.5%, >8.5%). The 95% Confidence Limits (CL) were calculated using asymptotic Wald method. Only positively adjudicated severe hypoglycemia and diabetic ketoacidosis were included in the analysis; Test type: Superiority — A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints were reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance <= 0.05; Percentage difference = 16.3, 95% CI 2-sided [9.17 to 23.43] — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; P-values were obtained from a CMH test stratified by the different levels of the randomization stratification factors of insulin delivery method (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%). The 95% CL were calculated using asymptotic Wald method; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance <= 0.05; Percentage difference = 17.2, 95% CI 2-sided [10.06 to 24.35] — Sotagliflozin 400 mg versus Placebo

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model. A negative change from baseline indicates a loss in body weight from baseline to Week 24.
Time Frame: Baseline to Week 24
Population: Analysis included participants from the mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 240 | 240 | 241
Kilograms (kg) | 0.11 (0.201) | -1.88 (0.200) | -2.47 (0.199)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -1.98, 95% CI 2-sided [-2.53 to -1.44], Standard Error of Mean 0.276 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM; Least squares mean difference = -2.58, 95% CI 2-sided [-3.12 to -2.04], Standard Error of Mean 0.276 — Sotagliflozin 400 mg versus Placebo

4. Secondary Outcome: Change From Baseline in Mean Daily Bolus Insulin Dose at Week 24
Description: The mean bolus insulin dose in international units/day (IU/day) for Week 24 was the average over the 3 to 5 days prior to the Week 24 visit. The Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post baseline values. A negative change from baseline indicated a reduction in the amount of bolus insulin used and a positive change from baseline indicated an increase in the amount of bolus insulin used between baseline and Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: IU/day
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 238 | 237 | 239
IU/day | -1.19 (0.635) | -4.38 (0.636) | -4.78 (0.634)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and Baseline mean daily bolus insulin dose-by-time interaction as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <=0.05; Least squares mean difference = -3.2, 95% CI 2-sided [-4.86 to -1.53], Standard Error of Mean 0.847 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -3.59, 95% CI 2-sided [-5.25 to -1.93], Standard Error of Mean 0.845 — Sotagliflozin 400 mg versus Placebo

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: The Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post baseline values. A negative change from baseline indicates a lower glucose level at Week 24 compared to baseline and a positive change from baseline indicates an increase in glucose level at Week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter (mg/dL)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 239 | 237 | 239
Milligram per deciliter (mg/dL) | 8.8 (3.95) | -12.8 (3.97) | -16.9 (3.96)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline Fasting Plasma Glucose-by-time interaction as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -21.6, 95% CI 2-sided [-32.2 to -11], Standard Error of Mean 5.38 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -25.7, 95% CI 2-sided [-36.2 to -15.1], Standard Error of Mean 5.37 — Sotagliflozin 400 mg versus Placebo

6. Secondary Outcome: Change From Baseline in Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score at Week 24
Description: The DTSQ instrument contains 8 items assessing overall treatment satisfaction, treatment convenience and flexibility, satisfaction with understanding of diabetes, willingness to continue present treatment and to recommend it to others, and frequency of unacceptably high and unacceptably low blood glucose levels. 6 items (1, 4, 5, 6, 7 and 8) (excluding perceived hyperglycemia and hypoglycemia items) were scored using a 7- point scale where 0=very dissatisfied to 6= very satisfied for a total possible score of 0 (very dissatisfied) to 36 (very satisfied), where higher scores indicate higher satisfaction from treatment. Two items (Q2 and 3), which were not included, measured perceived hyperglycemia and hypoglycemia, respectively. The baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post baseline values. A positive change from baseline indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 228 | 229 | 240
Score on a scale | -0.1 (0.28) | 1.9 (0.28) | 1.6 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline DTSQs total score-by-time interaction as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = 2, 95% CI 2-sided [1.3 to 2.7], Standard Error of Mean 0.37 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, MMRM — Threshold for significance <= 0.05; Least squares mean difference = 1.7, 95% CI 2-sided [1 to 2.4], Standard Error of Mean 0.36 — Sotagliflozin 400 mg versus Placebo

7. Secondary Outcome: Change From Baseline in 2-Item Diabetes Distress Screen 2 (DDS2) Score at Week 24
Description: DDS2 is a 2-item diabetes distress screening instrument where participants rated the degree to which the following items caused distress: (1) feeling overwhelmed by the demands of living with diabetes, and (2) feeling that I am often failing with my diabetes regimen using a 6-point scale: where 1=no distress to 6=severe distress for a total possible score of 2 to 12. LS means were obtained from MMRM model including all available post baseline values. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 232 | 232 | 243
Score on a scale | 0.0 (0.12) | -0.3 (0.12) | -0.4 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<= 8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline DDS2 total score-by-time interaction as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.025, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -0.3, 95% CI 2-sided [-0.6 to 0], Standard Error of Mean 0.15 — Sotagliflozin 200 mg versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; LS means and p-values were obtained from MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week -2 A1C (<=8.5%, >8.5%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline DDS2 total score-by-time interaction as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.003, MMRM — Threshold for significance <= 0.05; Least squares mean difference = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.15 — Sotagliflozin 400 mg versus Placebo

8. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model. A negative percent change from baseline indicates a loss in body weight from baseline to Week 24.
Time Frame: Baseline to Week 24
Population: Analysis included participants from the mITT population, including all available post baseline values. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 240 | 240 | 241
Percent change | 0.10 (0.245) | -2.38 (0.245) | -2.99 (0.244)

ADVERSE EVENTS:
Time Frame: First dose and up to 30 days after the last dose of double-blind study treatment. Some Adverse events may have been attributed to the long-term effects of study drug; included even if the onset was >30 days after the last dose of study drug (up to 393 days).
Description: Safety Population consisted of all randomly assigned participants treated with at least 1 dose of study drug, analyzed according to their actual treatment received.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 2/258 | 0/261 | 0/263
Serious Adverse Events (participants affected / at risk) | 17/258 | 26/261 | 21/263
Other Adverse Events (participants affected / at risk) | 46/258 | 52/261 | 64/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=258) | Sotagliflozin 200 mg (N=261) | Sotagliflozin 400 mg (N=263)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Prepyloric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Goiter (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 7 (7) | 12 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ecthyma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=258) | Sotagliflozin 200 mg (N=261) | Sotagliflozin 400 mg (N=263)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 12 (18) | 20 (29)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 40 (58) | 44 (60) | 49 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.